CLINICAL TRIAL: NCT05597735
Title: A Phase III, Multi-country, Randomized, Placebo-controlled, Double-blinded Trial to Assess the Efficacy and Safety of Tecovirimat Antiviral Treatment for Patients With Monkeypox Virus Disease
Brief Title: Assessment of the Efficacy and Safety of Tecovirimat in Patients With Monkeypox Virus Disease
Acronym: UNITY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University Hospital, Geneva (Other); Oswaldo Cruz Foundation (Other); Fundacion Huesped, Buenos Aires, Argentina (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-01579
Record Dates: First submitted 2022-10-27; First posted 2022-10-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-10

CONDITIONS: Monkeypox; Mpox
Keywords: Tecovirimat; Antiviral agent
MeSH Terms: conditions — Mpox, Monkeypox | interventions — tecovirimat

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, Double-blinded Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tecovirimat (Experimental)
  Interventions: Drug: Tecovirimat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tecovirimat — The experimental intervention is tecovirimat, available as immediate-release capsules containing tecovirimat monohydrate, equivalent to 200 mg of tecovirimat. The route of administration of tecovirimat is oral. Tecovirimat treatment will be initiated as soon as possible after diagnosis.
  The international recommended doses will be followed:
  * 25 kg to less than 40 kg: 400 mg (two tecovirimat 200 mg capsules) every 12 hours for 14 consecutive days.
  * 40 kg and above: 600 mg (three tecovirimat 200 mg capsules) every 12 hours for 14 consecutive days.
  Arms: Tecovirimat
Drug: Placebo — The control intervention is a placebo and its route of administration will be identical to the experimental intervention administration to allow treatment arm blinding.
  Arms: Placebo

SUMMARY:
The overall purpose of this study is to evaluate whether tecovirimat is an efficient and safe antiviral in the treatment of monkeypox in adults and adolescents (14 years old and older).

The primary objective is to evaluate the clinical efficacy, as assessed by time to all visible lesion(s) resolution, of tecovirimat treatment + Standard of Care (SOC) compared to placebo + SOC for patients with monkeypox.

The secondary objective is to evaluate the clinical efficacy, as assessed by mortality, hospitalization, complications, duration of symptoms and virological shedding, and the safety of tecovirimat treatment + SOC compared to placebo + SOC in patients with monkeypox.

DETAILED DESCRIPTION:
The study presented here is the Swiss-Brazil co-sponsored adaptation of the UNITY trial based on the WHO core protocol. It has an original governance to better respond to public health priorities, each country being its own sponsor, allowing for an easier scale-up of the trial and local adaptations of the protocol.

Background and rationale:

Monkeypox is an emerging viral zoonosis caused by a virus of the same name that is closely related to smallpox. It is usually endemic in central and West Africa but since May 2022, the virus has rapidly disseminated to Europe, North and South America, Africa and Australia, and has predominantly affected gay, bisexual and other men who have sex with men (MSM) with multiple partners. On 23 July 2022, the World Health Organization (WHO) declared that the monkeypox outbreak was an international public health emergency. In particular, the WHO called for the use of antivirals for the treatment of monkeypox cases. This declaration must therefore be translated not only into extraordinary public health measures but also as a call for greater investment in research.

This study proposal is a national adaptation for Switzerland and Brazil based on the 'CORE protocol' developed by the WHO. The research team would like to emphasize that this randomized trial is international in scope. Thus, they are joining forces to achieve a more effective and rapid response to important questions, with a harmonized follow-up and in a time frame that can be useful to the patients the medical staff have been caring for since the very beginning of this epidemic. Candidate antivirals are already available for testing in monkeypox. The first studied treatment in this adaptative trial is the antiviral tecovirimat. Tecovirimat (TPOXX®, SIGA Technologies Inc.) is a treatment for smallpox, monkeypox and cowpox. Tecovirimat is approved by the European Medicine Agency (EMA) for this indication for adults and children weighing at least 13 kg, as well as by the United States Food and Drugs Administration (FDA) under expanded access investigational new drug protocol, but it is not yet approved in Switzerland and Brazil.

Objectives:

This study aims to evaluate whether tecovirimat is an efficient and safe antiviral in the treatment of monkeypox in adults and adolescents (14 years old and over).

The primary objective is to evaluate the clinical efficacy of tecovirimat treatment + standard of care (SOC) compared to placebo + SOC for patients with monkeypox as assessed by time to visible lesion(s) resolution. The secondary objectives are to evaluate the clinical efficacy and safety of tecovirimat treatment + SOC compared to placebo + SOC in patients with monkeypox as assessed by mortality, hospitalization, complications, duration of symptoms and virological shedding.

Methods:

This study will include adult and adolescent patients aged ≥14 years with a confirmed or highly suspected monkeypox virus infection and with at least one visible active skin or mucosal lesion. Individuals with a known hypersensitivity to tecovirimat, who are taking medications which cannot be interrupted and for which a major interaction has been described or who, in the judgement of the investigator, will be at significantly increased risk as a result of participation in the study will not be included. Randomization will be in a ratio of 1:1 to either tecovirimat treatment combined with SOC or to placebo combined with SOC. All participants will be followed-up until day 29 and additionally at day 60 for those who accept this last optional follow-up visit.

Outcome:

The primary outcome is the time for all visible lesions (skin, mucosal) to heal with a new fresh layer of skin re-epithelialization (i.e. resurfacing of a wound with a new epithelium layer).

Expected results:

The hypothesis is that prompt oral treatment with tecovirimat will result in a reduction of the duration of illness in patients with monkeypox that may correlate with the duration of contagiousness. It is expected that tecovirimat will be well tolerated and acceptable for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults and adolescents (14 years old and older) with laboratory-confirmed (PCR if available) or highly suspected monkeypox virus infection of any duration
* At least one visible active skin or mucosal lesion
* Reachable via smartphone (for video calls) for outpatient participants
* Signed informed consent

Exclusion Criteria:

* Current or planned use of another investigational drug at any point during study participation.
* Ongoing treatment which cannot be interrupted and for which a major interaction has been described with tecovirimat
* Patients who, in the judgement of the investigator, will be at significantly increased risk as a result of participation in the study (for example: if the investigator judges that an antiviral treatment is indicated in the framework of compassionate therapeutic access in Switzerland).
* Hypersensitivity to tecovirimat

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Time to all visible lesion(s) resolution | 28 days
  Time for all visible lesions (skin, mucosal) to heal with a new fresh layer of skin re-epithelialization (i.e resurfacing of a wound with a new epithelium layer). For skin lesions, typically this means the lesion has scabbed, desquamated and new layer of skin has been formed. For mucosal lesions, the phase of scabbing and desquamation is absent, and healing with new layer of skin ensues.

SECONDARY OUTCOMES:
All-cause mortality within the first 28 days (applied to all patients) | 28 days
  All-cause mortality is more reliably measured than monkeypox-specific mortality. It is easy to measure and is reliable.
All-cause unplanned admission to hospital within first 28 days (applies to outpatients) | 28 days
  Most patients will be managed at home or in community and this outcome is an important patient-centered and health system outcome. All-cause is easier to measure than monkeypox specific and will ease data burden.
Occurrence of patients with a complication within first 28 days (applies to all patients who did not already have a complication at baseline) | 28 days
  Complications include secondary bacterial skin infection (cellulitis, abscess, necrotizing fasciitis, need for antibiotics), severe pain, ocular impairment (e.g. keratitis), neurologic impairment (e.g. encephalitis) or mental health disturbance, confusion, cardiac impairment (e.g. cardiomyopathy, myocarditis), severe dehydration, and genitourinary complications as urinary retention. Progression to complications is an important patient-centered outcome and an important health system outcome to prepare and anticipate clinical services for monkeypox cases. It is easy to measure, as long as definitions are clear, and the relevant staff is trained. Complications will be differentiated based on drug-related complications and disease-related complications.
Time to resolution of symptoms and signs within first 28 days (applies to all patients) | 28 days
  Symptoms include fatigue, malaise, nausea, vomiting, abdominal pain, anorexia, cough, dysphagia, odynophagia, fever, headache, oral pain, pain with urination, rectal/anal pain. Signs include lymphadenopathy, ocular lesions, pharyngitis, urethritis, and proctitis. Collection of symptoms and signs can be useful to understand the clinical characterization.
Viral clearance up to 28 days after randomization | 28 days
  Occurrence of negative oropharyngeal , rectal swab, and skin swab PCR results, respectively, 7, 14, 21 days and 28 days after randomization. Viral clearance assessment is important to evaluate whether treatment is also a route for reducing transmission.
Frequency of adverse events (AEs) and serious adverse events (SAEs) for specific therapeutics (applies to all patients) | 60 days
  The collection of standardized data of adverse events is of importance in order to increase the understanding of safety and tolerability of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yazdan Yazdapanah, Pr., Study Director — ANRS, Emerging Infectious Diseases
Locations (12):
- Fundación Huésped, Buenos Aires, Argentina
- Brazil (7):
  - Faculty of Medicine, Federal University of Minas Gerais, Belo Horizonte
  - Evandro Chagas National Institute of Infectious Diseases-Oswaldo Cruz Foundation-FIOCRUZ, Rio de Janeiro
  - Federal Hospital for State Employees, Rio de Janeiro
  - Nova Iguaçu General Hospital, Rio de Janeiro
  - University Hospital Prof. Edgard Santos, Salvador
  - Emílio Ribas Institute of Infectious Diseases, São Paulo
  - STD/AIDS Reference and Training Center, São Paulo
- Switzerland (4):
  - Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva
  - Pr Alexandra Calmy, Geneva, Canton of Geneva
  - CHUV, Lausanne, Canton of Vaud
  - Zürich checkpoint, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thornhill JP, Barkati S, Walmsley S, Rockstroh J, Antinori A, Harrison LB, Palich R, Nori A, Reeves I, Habibi MS, Apea V, Boesecke C, Vandekerckhove L, Yakubovsky M, Sendagorta E, Blanco JL, Florence E, Moschese D, Maltez FM, Goorhuis A, Pourcher V, Migaud P, Noe S, Pintado C, Maggi F, Hansen AE, Hoffmann C, Lezama JI, Mussini C, Cattelan A, Makofane K, Tan D, Nozza S, Nemeth J, Klein MB, Orkin CM; SHARE-net Clinical Group. Monkeypox Virus Infection in Humans across 16 Countries - April-June 2022. N Engl J Med. 2022 Aug 25;387(8):679-691. doi: 10.1056/NEJMoa2207323. Epub 2022 Jul 21. PMID 35866746
- [Background] Girometti N, Byrne R, Bracchi M, Heskin J, McOwan A, Tittle V, Gedela K, Scott C, Patel S, Gohil J, Nugent D, Suchak T, Dickinson M, Feeney M, Mora-Peris B, Stegmann K, Plaha K, Davies G, Moore LSP, Mughal N, Asboe D, Boffito M, Jones R, Whitlock G. Demographic and clinical characteristics of confirmed human monkeypox virus cases in individuals attending a sexual health centre in London, UK: an observational analysis. Lancet Infect Dis. 2022 Sep;22(9):1321-1328. doi: 10.1016/S1473-3099(22)00411-X. Epub 2022 Jul 1. PMID 35785793
- [Background] Siegrist EA, Sassine J. Antivirals With Activity Against Mpox: A Clinically Oriented Review. Clin Infect Dis. 2023 Jan 6;76(1):155-164. doi: 10.1093/cid/ciac622. PMID 35904001
- [Background] Smith SK, Self J, Weiss S, Carroll D, Braden Z, Regnery RL, Davidson W, Jordan R, Hruby DE, Damon IK. Effective antiviral treatment of systemic orthopoxvirus disease: ST-246 treatment of prairie dogs infected with monkeypox virus. J Virol. 2011 Sep;85(17):9176-87. doi: 10.1128/JVI.02173-10. Epub 2011 Jun 22. PMID 21697474
- [Background] O'Laughlin K, Tobolowsky FA, Elmor R, Overton R, O'Connor SM, Damon IK, Petersen BW, Rao AK, Chatham-Stephens K, Yu P, Yu Y; CDC Monkeypox Tecovirimat Data Abstraction Team. Clinical Use of Tecovirimat (Tpoxx) for Treatment of Monkeypox Under an Investigational New Drug Protocol - United States, May-August 2022. MMWR Morb Mortal Wkly Rep. 2022 Sep 16;71(37):1190-1195. doi: 10.15585/mmwr.mm7137e1. PMID 36107794
- [Background] Desai AN, Thompson GR 3rd, Neumeister SM, Arutyunova AM, Trigg K, Cohen SH. Compassionate Use of Tecovirimat for the Treatment of Monkeypox Infection. JAMA. 2022 Oct 4;328(13):1348-1350. doi: 10.1001/jama.2022.15336. PMID 35994281
- [Background] Adler H, Gould S, Hine P, Snell LB, Wong W, Houlihan CF, Osborne JC, Rampling T, Beadsworth MB, Duncan CJ, Dunning J, Fletcher TE, Hunter ER, Jacobs M, Khoo SH, Newsholme W, Porter D, Porter RJ, Ratcliffe L, Schmid ML, Semple MG, Tunbridge AJ, Wingfield T, Price NM; NHS England High Consequence Infectious Diseases (Airborne) Network. Clinical features and management of human monkeypox: a retrospective observational study in the UK. Lancet Infect Dis. 2022 Aug;22(8):1153-1162. doi: 10.1016/S1473-3099(22)00228-6. Epub 2022 May 24. PMID 35623380
- [Background] Carvalho T. The unknown efficacy of tecovirimat against monkeypox. Nat Med. 2022 Nov;28(11):2224-2225. doi: 10.1038/d41591-022-00094-0. No abstract available. PMID 36100750
- [Background] Merchlinsky M, Albright A, Olson V, Schiltz H, Merkeley T, Hughes C, Petersen B, Challberg M. The development and approval of tecoviromat (TPOXX(R)), the first antiviral against smallpox. Antiviral Res. 2019 Aug;168:168-174. doi: 10.1016/j.antiviral.2019.06.005. Epub 2019 Jun 7. PMID 31181284
- See also: Second meeting of the International Health Regulations (2005) (IHR) Emergency Committee regarding the multi-country outbreak of monkeypox — https://www.who.int/news/item/23-07-2022-second-meeting-of-the-international-health-regulations-(2005)-(ihr)-emergency-committee-regarding-the-multi-country-outbreak-of-monkeypox
- See also: CORE PROTOCOL - An international adaptive multi-country randomized,placebo-controlled, double-blinded trial of the safety and efficacy of treatments for patients with monkeypox virus disease — https://www.who.int/publications/m/item/core-protocol---an-international-adaptive-multi-country-randomized-placebo-controlled--double-blinded-trial-of-the-safety-and-efficacy-of-treatments-for-patients-with-monkeypox-virus-disease